CLINICAL TRIAL: NCT07204405
Title: Haemorrhage From Severe Neck and Facial Injuries - Characteristics, Management and Outcomes
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Hedberg, MD, PhD, Karolinska Institutet
Other Study IDs: K 2025-7172
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Trauma (Including Fractures); Facial Bones Fracture; Neck Injuries
Keywords: Facial injury; Neck injury; Trauma; Bleeding
MeSH Terms: conditions — Wounds and Injuries; Neck Injuries; Facial Injuries; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive observational study of trauma patients admitted to the Trauma Unit at the Karolinska University Hospital Solna, Stockholm, Sweden. Data will be collected from the Karolinska Trauma Registry for all patients from 2015 to 2024. A more detailed dataset will be extracted from the Trauma Registry for all patients with serious facial or neck injuries. For those patients, data will also manually be extracted from their clinical records.

DETAILED DESCRIPTION:
Data will be collected from the Karolinska Trauma Registry for all patients from 2015 to 2024. A more detailed dataset will be extracted from the Trauma Registry for all patients with an Abbreviated Injury Scale (AIS) severity score of ≥ 3 for facial or neck injuries. Data will include demographics, injury mechanism, injury type, physiology, treatment and outcome. For those patients with a severe facial or neck injury, data will also manually be extracted from their clinical records regarding prehospital details, initial physiology, injury type, treatment and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the Karolinska Trauma Registry

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in the Karolinska Trauma Registry. Those with an AIS>2 for neck or facial injury will be studied in more detail.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Death from bleeding | 30 days
  Death from bleeding within 30 days.

IPD SHARING:
Plan to Share IPD: No